CLINICAL TRIAL: NCT02275468
Title: Fu-zheng-qu-zhuo Oral Liquid Combined With Integrated Therapy Improves Renal Function in Patients of Chronic Kidney Disease Stage 3 and 4，a Randomized Placebo-Control Clinical Trial
Brief Title: Fu-zheng-qu-zhuo Oral Liquid Improves Renal Function in Patients of CKD Stage 3 and 4
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: Fangshan Hospital of Traditional Chinese Medicine, (Other); Peking University First Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SF-2009-Ⅲ-01
Record Dates: First submitted 2014-10-23; First posted 2014-10-27 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2014-10

CONDITIONS: Stage 3 Chronic Kidney Disease; Stage 4 Chronic Kidney Disease
Keywords: Chronic Kidney Disease; eGFR slope; Herbal medicine Fu-zheng-qu-zhuo Oral liquid
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — fu-zheng-qu-zhuo; Fluid Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (Placebo Comparator): Patients of Control Group received FZQZ-Placebo 20ml every time, and three times a day combined with integrated therapy.The integrated therapy was as follows: (1)low-protein dietary with sufficient calorie supply.(2) Anti-hypertensive agents to achieve a systolic blood pressure of less than 140 mm Hg and a diastolic blood pressure of less than 90 mmHg.(3)Anti-hyperlipidemic agentsas necessary to achieve low-density lipoprotein cholesterol（LDL-CH）less than 2.6mmol/L and triglycerides less than1.7mmol/L.（4）Patients with Diabetes Mellitus received insulin or oral hypoglycemic agents to achieve HbA1c 6.5～8.0%. (5)Received Sodium Bicarbonate as necessary to achieve serum HCO3-≥22mmol/L.(6) Received ferrous succinate, folic acid, and erythropoietin to achieve HB 90~110g/L.
- Fu-zheng-qu-zhuo oral liquid Group (Experimental): Patients of FZQZ Group received Fu-zheng-qu-zhuo (FZQZ) oral liquid 20ml every time, and three times a day combined with integrated therapy. The integrated therapy was same to Control Group.
  Interventions: Drug: Fu-zheng-qu-zhuo (FZQZ) oral liquid

INTERVENTIONS:
Drug: Fu-zheng-qu-zhuo (FZQZ) oral liquid — FZQZ oral liquid is a herbal medicine, composed of astragalus, angelica root, rhubarb, etc, with the effect of reinforcing Qi and activating blood, dissolving dampness and downbearing turbid.
  Other Names: FZQZ oral liquid
  Arms: Fu-zheng-qu-zhuo oral liquid Group

SUMMARY:
a prospective, multicenter (outpatient clinics of the three participating hospitals in Beijing), double blinded and randomized placebo-controlled study.

The study consisted of a 2-week run-in period and a 12-month treatment period.

ELIGIBILITY:
Inclusion Criteria:

(1) Signed informed consent and aged from 18 to 75 years old. (2) Chronic renal diseases with Glomerular Filtration Rate (GFR) estimated using the CKD Epidemiology Collaboration (CKD-EPI) equation between 15 and 59 ml/min per 1.73 m2 on at least 2 dates separated by at least 90 days but no more than 6 month (the CKD defining window period). (3)Not received other TCM treatment for at least 2 weeks.

Exclusion Criteria:

(1) 50% increase in serum creatinine occurring within 2 month before screening. (2) Immediate need for dialysis. (3) Myocardial infarction or cerebrovascular accident in the 6 month preceding the trial. (4) Connective-tissue disease, obstructive uropathy and renal transplantation. (5) Patients with severe disease in other organs or cancer, psychotic diseases, and active tuberculosis. (6) Treatment with corticosteroid and immunosuppressive agents in recent 3 month. Hemoglobin (Hb) less than 80 g/L. (7) Diabetes Mellitus with uncontrolled Blood Sugar ( glycated hemoglobin （HbA1c） >8.0%). (8) Enrolled in other trials. (9) Women in pregnancy or lactation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2010-06; Primary Completion 2013-05 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
composite end point | 12 month after the treatmnet and 3 years of the follow up time
  end stage renal disease (defined by the need for long-term dialysis or renal transplantation, or eGFR<15ml/min) and all cause of death

SECONDARY OUTCOMES:
the slope of the eGFR versus observation time | 12 month after the treatment
  the decline of eGFR per-year

CONTACTS AND LOCATIONS:
Overall Officials: Jie Wang, Study Chair — Guang anmen Hospital, China Academy of Chinese Medical Sciences
Locations (3):
- China (3):
  - Guang anmen Hospital, China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality
  - Fangshan Hospital of Traditional Chinese Medicine, Beijing, Beijing Municipality
  - Guang'an Men Hospital South, Beijing